CLINICAL TRIAL: NCT07167797
Title: Evaluation of the Role of Vitamin D in Reducing the Severity and Duration of Rotavirus Infection in Iraqi Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Fadia Thamir Ahmed, Lecturer/ College of Pharmacy/ University of Baghdad, University of Baghdad
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1969
Record Dates: First submitted 2025-08-21; First posted 2025-09-11 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Rotaviral Gastroenteritis
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (control): received standard treatment which include rehydration therapy and antipyretic the (Placebo Comparator): Group I (control): will receive standard treatment which include rehydration therapy and antipyretic therapy
  Interventions: Drug: Standard treatment for rotavirus
- Group II (Treatment) group: received vitamin D single oral dose 300000 IU for age < 1 year and dose (Experimental): Group II (Treatment) group: received vitamin D single oral dose 100000 IU for age < 1 year and dose of 300000IU for age> 1 year in addition to standard treatment. The study lasted 6 months, with follow-ups at 7-10 days
  Interventions: Dietary Supplement: Vitamin D (Cholecalciferol )

INTERVENTIONS:
Dietary Supplement: Vitamin D (Cholecalciferol ) — Group II (Treatment) group: received vitamin D single oral dose 100000 IU for age < 1 year and dose of 300000IU for age> 1 year in addition to standard treatment
  Arms: Group II (Treatment) group: received vitamin D single oral dose 300000 IU for age < 1 year and dose
Drug: Standard treatment for rotavirus — Standard treatment for rotavirus which includes rehydration therapy and antipyretic therapy including sodium chloride fluid and paracetamol infusion
  Arms: Group I (control): received standard treatment which include rehydration therapy and antipyretic the

SUMMARY:
The aim of this study is to evaluate the effect of vitamin D supplementation on the clinical outcomes including duration and severity of rotavirus-induced gastroenteritis in children that will be admitted to the hospital. And to evaluate the anti-inflammatory effect of vitamin D on the pediatrics with rotavirus gastroenteritis by measuring inflammatory markers such as C-reactive protein (CRP), neutrophil to lymphocyte ratio (NLR), platelet to lymphocytes ratio (PLR), lymphocytes to monocytes ratio (LMR) and mean platelet volume MPV.

DETAILED DESCRIPTION:
Evaluation of effect of vitamin D supplementation on the clinical outcomes including duration and severity of rotavirus-induced gastroenteritis in children that will be admitted to the hospital. And to evaluate the anti-inflammatory effect of vitamin D on the pediatrics with rotavirus gastroenteritis by measuring inflammatory markers such as C-reactive protein (CRP), neutrophil to lymphocyte ratio (NLR), platelet to lymphocytes ratio (PLR), lymphocytes to monocytes ratio (LMR) and mean platelet volume MPV.

ELIGIBILITY:
Inclusion Criteria:

1. Children with confirmed rotavirus infection by rotavirus stool examination by rotavirus rapid test from CerTest BIOTEC company in Spain.
2. Serum vitamin D levels indicating deficiency (below 20 ng/mL)

Exclusion Criteria:

1. Children with other major infections, severe dehydration or underlying health conditions.
2. Children with current vitamin D supplementation.

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-12-06 (Actual)

PRIMARY OUTCOMES:
Severity of diarrhea | 7 days
  severity of diarrhea will be measured by frequency of daily bowel movement
Duration of diarrhea | 7 days
  Duration of diarrhea will be measured by days
Severity of vomiting | 7 days
  Severity of vomiting will be measured by frequency of vomiting per day
Duration of vomiting | 7 days
  Duration of vomiting will be measured by days
Hydration state | 7 days
  Hydration state will be measured by score (1 fore well hydrated,2 for mild dehydration, 3 for moderate dehydration and 4 for severe dehydration)
Temperature | 7 days
  Temperature will be measured by nominal scale (1 for febrile and 0 fir afebrile patient)

SECONDARY OUTCOMES:
Measuring LMR at admission, after 4 days and after 7 days both groups. | 7 days
  Measuring LMR will be done by getting ratios of blood cells from CBC test
C reactive protein (CRP) | 7 days
  CRP will be measured in mg/dl by CRP agglutination test
Mean platelet volume (MPV) | 7 days
  Mean platelet volume (MPV) will be measured in femtoliter (fL)
Measuring NLR at admission, after 4 days and after 7 days both groups. | 7 days
  Measuring NLR at admission, after 4 days and after 7 days both groups.
Measuring PLR at admission, after 4 days and after 7 days both groups. | 7 days
  Measuring PLR at admission, after 4 days and after 7 days both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- AL Kadhimia pediatric hospital, Baghdad, Baghdad Governorate, Iraq

IPD SHARING:
Plan to Share IPD: Yes
Participant data such as clinical outcomes, laboratory data and demographic data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: in March 2026 and will be always available
Access Criteria: Researchers will be able to access data from open access journal
URL: https://pharmacia.pensoft.net